CLINICAL TRIAL: NCT06865924
Title: Colangioids to Define the Genetic Factors Involved in Atypical Primary Sclerosing Cholangitis
Acronym: CILIA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Valenti:, Principal Investigation, Medical Doctor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CILIA
Record Dates: First submitted 2025-02-19; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: PSC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behaviour of the genetic variants involved in ciliopathies. (Experimental): Study of the onset and progression of aPSC by analyzing in three-dimensional models called assembloids:
  * Morphology of primary eyelashes
  * Differentiation of cholangiocytes
  * Activation of fibrogenesis
  * Infiltration of immune cells
  Interventions: Other: Use of assembloids as in vitro models to test new pharmacological approaches

INTERVENTIONS:
Other: Use of assembloids as in vitro models to test new pharmacological approaches — Using extracellular vesicles containing the CRISPR/Cas9 genome editing system that by faithfully reproducing the in vivo part will allow a more faithful response than the use of conventional 2D model, organoids or animal model.

SUMMARY:
Primary sclerosing cholangitis (PSC) is a rare, progressive and often fatal disease of the intrahepatic or extrahepatic bile ducts, with an estimated prevalence in Western countries of 1/10,000. Biliary disease in PSC is represented by cholestasis, chronic inflammation of the bile ducts, the small tubes through which bile passes, progressive concentric fibrosis around the bile ducts2. This results in an obstruction to the passage of bile, which can lead to the development of cirrhosis with complications related to portal hypertension, cholangitis and often progress to bile duct cancer (cholangiocarcinoma). The only curative therapy in patients with PSC is liver transplantation, since no drug has been shown to be effective in preventing disease progression. The etiology is most likely multifactorial immune-mediated, where the onset of PSC is triggered by environmental factors in a genetically susceptible host2Genome-wide association studies (GWAS) have identified variations at the human leukocyte antigen (HLA) complex on chromosome 6 and several other loci, but these explain only a small part of the heritability of PSC. In most cases, PSC occurs in men in their 30s and 40s who have inflammatory bowel disease (IBD) suggesting a key role of altered intestinal permeability and inflammation. However, approximately 30% of patients do not present colonic inflammation, which is consistent with the heterogeneity of the disease. Preliminary data obtained in our laboratory analyzing a cohort of Italian individuals with atypical PSC (aPSC), identified a suggestive enrichment of rare variants in genes involved in cilia morphogenesis (CEP120 and AHI1). These data are consistent with previous findings, showing the correlation between gene variants involved in ciliopathies, including the DCDC26 gene, and chronic cholestatic disorders that can mimic PSC. Primary cilia are organelles present on the outer membrane of ductal cells, called cholangiocytes. These organelles function as antennas that detect stimuli from bile and transmit information to cells by regulating various signaling pathways involved in secretion, proliferation and apoptosis. Therefore, the alteration of primary cilia plays an important role in the de-differentiation of cholangiocytes and therefore in the development of cholangiopathies, in the invasion of inflammatory cells and in the fibrotic process. However, to date little is known about the contribution of genetic variants to the severity and progression of PSC, perhaps also due to the lack of a reliable model of bile duct. Recently, three-dimensional cell cultures, called organoids, have been proposed as a revolutionary tool in the field of cell biology, as they are able to mimic the corresponding organ in vivo.Organoids can be derived from either induced pluripotent stem cells (iPSCs) or tissue-resident adult stem cells. Compared to conventional 2D cultures and animal models, organoids allow to reproduce the genetic background of the patient in the model, recapitulating in vitro structures and functions similar to in vivo tissues. For this reason, organoids have been exploited in different applications, including drug discovery and testing, precision medicine and cell therapy 9311. However, organoids still show several limitations to model liver diseases. Indeed, they are only able to recapitulate the hepatic epithelial component, cholangiocytes and/or hepatocytes and above all they lack the 3D hepatic microenvironment, such as stromal and immune cells, which play an important role in the pathogenesis of several liver diseases. The present study is part of a project funded by the Regional Foundation for Biomedical Research (FRRB) whose general objective is to generate three-dimensional models of primary sclerosing cholangitis (PSC), called assemblyloids, and to study the cellular and molecular mechanisms through which genetic variants associated with genes involved in ciliopathies accelerate the progression of PSC. Our hypothesis is that the loss of function of cilia in cholangiocytes may represent a link between cellular senescence, development of inflammation, fibrosis and finally liver cancer. The variants related to ciliopathies could lead to an incomplete maturation of cholangiocytes with consequent malfunction that can therefore lead to a chronic inflammation of ductal cells and therefore to a persistent and uncontrolled activation of stromal cells and infiltration of immune cells. Furthermore, the generation of assemblyloids capable of reproducing native tissue as faithfully as possible will provide a new in vitro model for testing new pharmacological approaches aimed at correcting genetic mutations for improved precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 90 years of age
* Of both sexes
* willingness to sign informed consent for the study; Additional criteria group 1
* Patients with a confirmed aPSC diagnosis Additional criteria group 2
* patients with suspected PSC liver biopsy candidates Additional criteria group 3
* Patients not affected by aPSC listed for the following procedures:
* Liver resection for hepatocellular or other hepatic lesions (including secondary effects from other cancers and benign focal lesions, which will result in healthy liver tissue);
* Post-transplant biopsies of healthy liver;
* cholecystectomies. Additional criteria group 4
* Patients previously genotyped in the study "Impact of complete exoma sequencing on clinical management of patient with non-alcoholic liver steatosis and cryptogenic liver disease project code RF-2016-02364358" results carrying gene variants associated with ciliopathies

Exclusion Criteria:

-Positive for chronic viral hepatitis (HCV-RNA and HBsAg).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The quantify the impact of genetic risk factors for PSC and the role genetic variants | 48 months
  The different inclusion criteria are able to identify the number of individuals at risk for PSC among patients. Understand the impact of individual genetic variants on PSC risk and rates variants associated with ciliopathies on aPSC phenotype within the variant carrier group compared to the non-carrier group.

SECONDARY OUTCOMES:
The quantify the impact of pharmacological tests on extracellular vesicles | 48 months
  The impact of genetic risk factors for PSC and their interaction will be realized by evaluating the extracellular vesicles of the CRISPR/Cas9 genome editing system to correct mutations involved in ciliopathies.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Milano, Italy

DOCUMENTS (1):
  • Study Protocol (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT06865924/Prot_000.pdf